CLINICAL TRIAL: NCT03260894
Title: A Randomized, Open-Label, Phase 3 Study to Evaluate Efficacy and Safety of Pembrolizumab (MK-3475) Plus Epacadostat vs Standard of Care (Sunitinib or Pazopanib) as First-Line Treatment for Locally Advanced or Metastatic Renal Cell Carcinoma (mRCC) (KEYNOTE-679/ECHO-302)
Brief Title: Pembrolizumab (MK-3475) Plus Epacadostat vs Standard of Care in mRCC (KEYNOTE-679/ECHO-302)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KEYNOTE-679/ECHO-302; 2024-512016-22-00 (Registry Identifier: EU CT Number); 2017-002259-26 (EudraCT Number)
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Results first posted 2019-09-10 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Renal Cell Carcinoma (RCC)
Keywords: Renal cell carcinoma; programmed cell death 1 (PD-1) inhibitor; indoleamine 2; 3-dioxygenase 1 (IDO1) inhibitor
MeSH Terms: conditions — Carcinoma, Renal Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; epacadostat; Sunitinib; pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Epacadostat (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Epacadostat
- SoC (Sunitinib or Pazopanib) (Active Comparator): Standard of care (SoC) (sunitinib or pazopanib monotherapy).
  Interventions: Drug: Sunitinib; Drug: Pazopanib

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg administered intravenously every 3 weeks.
  Other Names: MK-3475
  Arms: Pembrolizumab + Epacadostat
Drug: Epacadostat — Epacadostat 100 mg administered orally twice daily.
  Other Names: INCB024360
  Arms: Pembrolizumab + Epacadostat
Drug: Sunitinib — Sunitinib 50 mg administered orally once daily; 4 weeks on, 2 weeks off for 6-wk cycle.
  Other Names: Sutent; SU11248
  Arms: SoC (Sunitinib or Pazopanib)
Drug: Pazopanib — Pazopanib 800 mg administered orally once daily.
  Other Names: Votrient
  Arms: SoC (Sunitinib or Pazopanib)

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of pembrolizumab plus epacadostat compared to sunitinib or pazopanib in participants with locally advanced/metastatic renal cell carcinoma (mRCC) with a clear cell component who have not received prior systemic therapy for their mRCC.

ELIGIBILITY:
Inclusion Criteria:

* Histologic confirmation of locally advanced or metastatic RCC with a clear-cell component with or without sarcomatoid features.
* Must not have received any prior systemic therapy for their mRCC.
* Measurable disease based on RECIST v1.1.
* Archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion as required.
* Karnofsky performance status ≥ 70%.
* Adequate organ function per protocol-defined criteria.

Exclusion Criteria:

* Use of protocol-defined prior/concomitant therapy.
* Currently receiving or has received an investigational treatment as part of a study of an investigational agent or has used an investigational device within 4 weeks before randomization.
* History of severe hypersensitivity reaction to study treatments or their excipients.
* Active autoimmune disease that has required systemic treatment in past 2 years.
* Known additional malignancy that has progressed or has required active treatment in the last 3 years.
* Known active central nervous system metastases and/or carcinomatous meningitis.
* History of (noninfectious) pneumonitis that required steroids or current pneumonitis.
* History or presence of an abnormal electrocardiogram that, in the investigator's opinion, is clinically meaningful.
* Significant cardiac event within 12 months before Cycle 1 Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2025-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Jones, MD, Study Director — Incyte Corporation
Locations (140):
- United States (25):
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Arizona Oncology Associates PC- HOPE, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UC Irvine Comprehensive Cancer Center/Chao Family Comprehensive Cancer Center, Orange, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Woodlands Medical Specialists, PA, Pensacola, Florida
  - Northside Hospital, Atlanta, Georgia
  - Atlanta Cancer Care - Conyers, Conyers, Georgia
  - Northwest Georgia Oncology Centers Pc, Marietta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Southeast Nebraska Hematology & Oncology Consultants, P.C., Lincoln, Nebraska
  - New York Oncology Hematology P.C, Albany, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - University of Tennessee Erlanger Oncology & Hematology, Chattanooga, Tennessee
  - The West Clinic, P.C., Germantown, Tennessee
  - US Oncology and Research, The Woodlands, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Oncology & Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Roanoke, Virginia
  - Shenandoah Oncology, P.C., Winchester, Virginia
- Australia (5):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Cabrini Health, Malvern, Victoria
  - Fiona Stanley Hospital, Murdoch
- Brazil (6):
  - Centro de pesquisa Porto Alegre, Porto Alegre, Florianopolis
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Sao Jose, São Paulo, São Paulo
  - Centro Avancado de Tratamento Oncologico - CENANTRON -, Belo Horizonte
  - Hospital de Clinicas de Porto Alegre, Porto Alegre
- Canada (6):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Kingston Health Sciences Centre - KGH Site, Kingston, Ontario
  - Sunnybrook Health Sciences, Odette Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-Universite Laval-Hotel Dieu de Quebec, Québec, Quebec
  - CIUSSS de la Mauricie-et-du-Centre-du-Quebec, Trois-Rivières, Quebec
- Chile (4):
  - Clinica Alemana de Osorno, Osorno, Los Lagos Region
  - Fundacion Arturo Lopez Perez FALP, Santiago
  - Pontificia Universidad Catolica de Chile, Santiago
  - Hospital Clinico Vina del Mar, Viña del Mar
- France (10):
  - Centre Antoine Lacassagne, Nice, Cedex 2
  - CHU Besancon - Hopital Jean Minjoz, Besançon
  - Hopital Saint Andre, Bordeaux
  - Centre Francois Baclesse, Caen
  - Hopital Prive Toulon Hyeres Sainte Marguerite, Hyères
  - Hopital Europeen Georges Pompidou, Paris
  - Hospices Civils de Lyon Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Clinique Sainte Anne, Strasbourg
  - CHU de Strasbourg - Nouvel Hopital Civil, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Germany (8):
  - Helios Klinikum Berlin Buch, Berlin
  - Universitaetsklinikum der Technischen Universitaet Dresden, Dresden
  - Universitaetsklinikum Essen, Essen
  - Universitaetsklinikum Frankfurt, Frankfurt am Main
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Magdeburg. Klinik fuer Urologie, Magdeburg
  - Universitaetsklinikum Tuebingen, Tübingen
- Hungary (6):
  - Orszagos Onkologiai Intezet, Budapest, Pest County
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg, Pozva
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet, Szolnok
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
- Ireland (2):
  - Adelaide & Meath Hospital, Dublin
  - University Hospital Waterford, Waterford
- Italy (6):
  - Medical Oncology Ospedale San Donato, Arezzo
  - Azienda Ospedaliera-Spedali Civili, Brescia
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - A.O. Cardarelli, Napoli
  - Policlinico San Matteo, Pavia
  - Azienda Ospedaliera San Camillo Forlanini, Roma
- Japan (14):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Nara Medical University Hospital, Kashihara, Nara
  - Kindai University Hospital, Sayama, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Yamaguchi University Hospital, Ube, Yamaguchi
  - Akita University Hospital, Akita
  - Kyushu University Hospital, Fukuoka
  - Niigata University Medical & Dental Hospital, Niigata
  - Toranomon Hospital, Tokyo
  - Nippon Medical School Hospital, Tokyo
  - Keio University Hospital, Tokyo
- Auckland City Hospital, Auckland, Grafton, New Zealand
- Norway (7):
  - Helse Bergen HF Haukeland sykehus, Bergen
  - Sykehuset Oestfold, Grålum
  - Sorlandet sykehus HF, Kristiansand
  - Akershus University Hospital, Lørenskog
  - Oslo universitetssykehus, Oslo
  - Universitetssykehuset i Nord Norge. Kreftavdelingen, Tromsø
  - St Olavs Hospital, Trondheim
- Russia (6):
  - Leningrad Regional Oncology Dispensary, Saint Petersburg, Leningrad Region, Vsevolozhsky District
  - Ivanovo regional oncology dispensary, Ivanovo
  - Russian Scientific Center of Roentgenoradiology, Moscow
  - Central Clinical Hospital with outpatient Clinic, Moscow
  - National Medical Research Radiology Centre, Moscow
  - Republican Clinical Oncology Dispensary of Republic of Bashkortostan, Ufa
- South Korea (4):
  - Chonnam National University Hwasun Hospital, Hwasun, Jeollanam-do
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (7):
  - Hospital Parc Tauli, Sabadell, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Instituto Valenciano de Oncologia, Valencia
- Taiwan (5):
  - Chang Gung Med Foundation. Kaohsiung Branch, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (7):
  - Baskent Universitesi Adana Dr. Turgut Noyan Uygulama ve Arastirma Merkezi, Adana
  - Ankara Numune Education and Research Hospital, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Istanbul Universitesi Onkoloji Enstitusu, Istanbul
  - Istanbul Medeniyet Universitesi Goztepe EAH, Istanbul
  - Ege Universitesi Tıp Fakultesi, Izmir
  - Namik Kemal Universitesi Tip Fakultesi, Tekirdağ
- Ukraine (5):
  - MI Kryviy Rih Center of Dnipropetrovsk Regional Council, Kryvyi Rih, Dnipropetrovsk Oblast
  - Dnipropetrovsk Regional Hospital n.a. I.I. Mechnikov, Dnipro
  - Dnipropetrovsk City Multidiscipline Clinical Hosp. 4 of DRC, Dnipro
  - MI Precarpathian Clinical Oncology Center, Ivano-Frankivsk
  - RMI Sumy Regional Clinical Oncology Dispensary, Sumy
- United Kingdom (6):
  - The Royal Marsden NHS Foundation Trust., Sutton, Surrey
  - Western General Hospital, Edinburgh
  - Beatson Institute of Cancer Research, Glasgow
  - Barts Health NHS Trust - St Bartholomew s Hospital, London
  - The Royal Marsden Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lara PN Jr, Villanueva L, Ibanez C, Erman M, Lee JL, Heinrich D, Lipatov ON, Gedye C, Gokmen E, Acevedo A, Semenov A, Park SH, Gafanov RA, Kose F, Jones M, Du X, Munteanu M, Perini R, Choueiri TK, Motzer RJ. A randomized, open-label, phase 3 trial of pembrolizumab plus epacadostat versus sunitinib or pazopanib as first-line treatment for metastatic renal cell carcinoma (KEYNOTE-679/ECHO-302). BMC Cancer. 2024 Jul 25;23(Suppl 1):1253. doi: 10.1186/s12885-023-10971-7. PMID 39054430

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 73 centers in 14 countries.
Groups:
- Pembrolizumab + Epacadostat: Pembrolizumab 200 mg administered intravenously every 3 weeks. Epacadostat 100 mg administered orally twice daily.
- SoC (Sunitinib or Pazopanib): Standard of care (SoC) (sunitinib or pazopanib monotherapy). Sunitinib 50 mg administered orally once daily;4 weeks on, 2 weeks off for 6-wk cycle. Pazopanib 800 mg administered orally once daily.
Period: Overall Study
Arm/Group | Pembrolizumab + Epacadostat | SoC (Sunitinib or Pazopanib)
Started | 64 | 65
Intention-to-Treat (ITT) | 64 | 65
All Subjects as Treated (ASaT) | 64 | 63
Completed | 18 | 15
Not Completed | 46 | 50
Not completed — Death | 6 | 8
Not completed — Withdrawal by Subject | 4 | 11
Not completed — On-going at clinical cut off date | 36 | 31

BASELINE CHARACTERISTICS:
Population: The Intention-to-Treat (ITT) population consisted of all randomized participants.
Groups:
- SoC (Sunitinib or Pazopanib): Standard of care (SoC) (sunitinib or pazopanib monotherapy). Sunitinib 50 mg administered orally once daily. Pazopanib 800 mg administered orally once daily.
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Epacadostat | SoC (Sunitinib or Pazopanib) | Total
Number analyzed (Participants) | 64 | 65 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (10.9) | 62.1 (10.6) | 62.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 15 | 35
  Male | 44 | 50 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 14 | 33
  Not Hispanic or Latino | 43 | 47 | 90
  Unknown or Not Reported | 2 | 4 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 1 | 0 | 1
  Asian | 10 | 9 | 19
  White | 53 | 56 | 109
ECOG Performance Scale [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) scale describes a patient's level of functioning in terms of their ability to care for themselves, activity, and ability. The scale is from 0 to 5; 0 - Fully active; 1 - Restricted in physically strenuous activity but ambulatory; 2- Ambulatory and capable of all selfcare but unable to carry out any work activities; 3- Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; 4 - Completely disabled; 5 - Dead.
  Participants
    0 | 41 | 35 | 76
    1 | 23 | 28 | 51
    2 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) of Pembrolizumab + Epacadostat Versus Standard of Care (SOC)
Description: ORR was defined as the percentage of participants who had complete response (CR) or partial response (PR) per RECIST v1.1 by investigator determination.
Time Frame: Minimum up to 6 months
Population: The Intention-to-Treat (ITT) population consisted of all randomized participants.
  Responses are based on Investigator assessments per RECIST 1.1 without confirmation using all scans up to the cutoff date 28FEB2019.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab + Epacadostat | SoC (Sunitinib or Pazopanib)
Number analyzed (Participants) | 64 | 65
percentage of participants
  Complete Response (CR): number analyzed (Participants) | 64 | 0
  Complete Response (CR) | 1.6 [0.0 to 8.4] |
  Partial Response (PR) | 29.7 [18.9 to 42.4] | 29.2 [18.6 to 41.8]
  Objective Response (CR+PR) | 31.3 [20.2 to 44.1] | 29.2 [18.6 to 41.8]

2. Secondary Outcome: Safety and Tolerability of Pembrolizumab + Epacadostat Versus SOC as Measured by the Number of Participants Experiencing Adverse Events (AEs)
Description: AE is defined as any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: Data reported from start of study to data cutoff 28-Feb-2019, up to 15 months.
Population: The All Subjects as Treated (ASaT) population was used for the safety analysis and consisted of all randomized participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Epacadostat | SoC (Sunitinib or Pazopanib)
Number analyzed (Participants) | 64 | 63
Participants | 64 | 63

3. Secondary Outcome: Safety and Tolerability of Pembrolizumab + Epacadostat Versus SOC as Measured by the Number of Participants Discontinuing Study Drug Due to AEs
Description: as for outcome 2
Time Frame: Data reported from start of study to data cutoff 28-Feb-2019, up to 15 months.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Epacadostat | SoC (Sunitinib or Pazopanib)
Number analyzed (Participants) | 64 | 63
Participants | 8 | 6

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were reported from start of study, up to 30 days after last dose and serious adverse events up to 90 days after last dose are included, up to 15 months
Description: The All Participants as Treated (APaT) population was used for the safety analysis and consisted of all randomized participants who received at least 1 dose of study treatment.
  All-Cause Mortality was based on the ITT population and consisted of all randomized participants.
  MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to the drug are excluded
Arm/Group | Pembrolizumab + Epacadostat | SoC (Sunitinib or Pazopanib)
All-Cause Mortality (participants affected / at risk) | 8/64 | 8/65
Serious Adverse Events (participants affected / at risk) | 18/64 | 15/63
Other Adverse Events (participants affected / at risk) | 61/64 | 61/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Epacadostat (N=64) | SoC (Sunitinib or Pazopanib) (N=63)
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2
Steroid diabetes (Metabolism and nutrition disorders) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Prostatomegaly (Reproductive system and breast disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab + Epacadostat (N=64) | SoC (Sunitinib or Pazopanib) (N=63)
Anaemia (Blood and lymphatic system disorders) | 10 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4
Hyperthyroidism (Endocrine disorders) | 5 | 2
Hypothyroidism (Endocrine disorders) | 9 | 12
Abdominal distension (Gastrointestinal disorders) | 4 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 9 | 3
Diarrhoea (Gastrointestinal disorders) | 13 | 30
Dry mouth (Gastrointestinal disorders) | 4 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 7
Nausea (Gastrointestinal disorders) | 22 | 20
Stomatitis (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 6 | 12
Asthenia (General disorders) | 2 | 6
Chest pain (General disorders) | 5 | 0
Fatigue (General disorders) | 12 | 15
Influenza like illness (General disorders) | 2 | 4
Oedema peripheral (General disorders) | 3 | 4
Pyrexia (General disorders) | 5 | 2
Alanine aminotransferase increased (Investigations) | 8 | 14
Amylase increased (Investigations) | 8 | 9
Aspartate aminotransferase increased (Investigations) | 4 | 16
Blood alkaline phosphatase increased (Investigations) | 6 | 9
Blood bilirubin increased (Investigations) | 1 | 9
Blood creatinine increased (Investigations) | 7 | 7
Blood lactate dehydrogenase increased (Investigations) | 1 | 5
Lipase increased (Investigations) | 6 | 9
Neutrophil count decreased (Investigations) | 0 | 4
Platelet count decreased (Investigations) | 1 | 6
Weight decreased (Investigations) | 7 | 2
Decreased appetite (Metabolism and nutrition disorders) | 10 | 12
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Dysgeusia (Nervous system disorders) | 1 | 8
Headache (Nervous system disorders) | 3 | 9
Insomnia (Psychiatric disorders) | 6 | 3
Haematuria (Renal and urinary disorders) | 4 | 3
Proteinuria (Renal and urinary disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 7
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 14
Pruritus (Skin and subcutaneous tissue disorders) | 16 | 1
Rash (Skin and subcutaneous tissue disorders) | 11 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 3
Hypertension (Vascular disorders) | 7 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-15): https://cdn.clinicaltrials.gov/large-docs/94/NCT03260894/Prot_SAP_000.pdf